CLINICAL TRIAL: NCT01956175
Title: A Single-centre, Double Blind, Randomised Controlled Clinical Trial to Evaluate the Effect of Electrical Pharyngeal Stimulation as a Treatment for Stroke-related Dysphagia in Tracheostomized Stroke Patients
Brief Title: Electrical Pharyngeal Stimulation for Dysphagia Therapy in Tracheostomized Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-580
Record Dates: First submitted 2013-09-24; First posted 2013-10-08 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Stroke; Dysphagia
Keywords: electrical pharyngeal stimulation; stroke-related dysphagia; tracheostomy; decannulation
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electrical pharyngeal stimulation (Experimental): Electrical pharyngeal stimulation once daily for 10 minutes on three consecutive days.
  Interventions: Device: Electrical pharyngeal stimulation
- Sham stimulation (Sham Comparator): Sham stimulation once daily for 10 minutes on three consecutive days. If the subject cannot be decannulated after three days of sham stimulation, another three days of real electrical pharyngeal stimulation will be delivered.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Electrical pharyngeal stimulation — Electrical pharyngeal stimulation via an intraluminal catheter (Phagenesis Ltd.) once daily for 10 minutes on three consecutive days. The intensity of the electrical stimulation is determined following the calculation of suitable sensory threshold, tailored to the individual participants. After determining the optimal stimulation intensity, 10 minutes of stimulation are delivered.
  Other Names: Phagenesis Limited, UK.; EPS1 device
  Arms: Electrical pharyngeal stimulation
Device: Sham stimulation — The intraluminal catheter (Phagenesis Ltd.) for electrical pharyngeal stimulation is placed. The intensity of the electrical stimulation is determined following the calculation of suitable sensory threshold, tailored to the individual participants. After the optimal stimulation intensity has been determined, no electrical stimulation is delivered.
  Arms: Sham stimulation

SUMMARY:
The purpose of this study is to evaluate whether electrical pharyngeal stimulation in addition to standard care can enhance short-term swallow recovery in tracheostomized dysphagic stroke patients and thereby facilitate earlier decannulation compared to sham treatment plus standard care.

DETAILED DESCRIPTION:
Readiness for decannulation is assessed after three days of either real or sham electrical pharyngeal stimulation. In case a patient cannot be decannulated at that time point, there is an open-label follow-up treatment phase, in which every patient in the sham treatment arm gets another three days of real electrical pharyngeal stimulation to not deprive any patient of a potentially beneficial treatment.

ELIGIBILITY:
Inclusion Criteria:

* severe dysphagia due to acute stroke
* completely weaned from mechanical ventilation
* impossibility of decannulation because of severe dysphagia with ongoing aspiration

Exclusion Criteria:

* preexisting dysphagia
* comorbidities that can possibly cause dysphagia
* psychiatric comorbidities
* pacemaker or other implanted electronic devices

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Readiness for decannulation | 3 days
  Difference in readiness for decannulation as assessed by a standardized fiberoptic endoscopic evaluation protocol after three days of treatment between real and sham treatment groups

SECONDARY OUTCOMES:
Functional Oral Intake Scale (FOIS) at discharge | until discharge
modified Rankin Scale (mRS) at discharge | until discharge
length of stay on ICU / in the hospital and time from stimulation to discharge | until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Dziewas, PhD, Principal Investigator — Department of Neurology, University of Muenster
Locations (1):
- Department of Neurology, University of Muenster, Münster, Muenster, Germany

REFERENCES:
- [Background] Warnecke T, Suntrup S, Teismann IK, Hamacher C, Oelenberg S, Dziewas R. Standardized endoscopic swallowing evaluation for tracheostomy decannulation in critically ill neurologic patients. Crit Care Med. 2013 Jul;41(7):1728-32. doi: 10.1097/CCM.0b013e31828a4626. PMID 23774336
- [Background] Fraser C, Power M, Hamdy S, Rothwell J, Hobday D, Hollander I, Tyrell P, Hobson A, Williams S, Thompson D. Driving plasticity in human adult motor cortex is associated with improved motor function after brain injury. Neuron. 2002 May 30;34(5):831-40. doi: 10.1016/s0896-6273(02)00705-5. PMID 12062028
- [Derived] Suntrup S, Marian T, Schroder JB, Suttrup I, Muhle P, Oelenberg S, Hamacher C, Minnerup J, Warnecke T, Dziewas R. Electrical pharyngeal stimulation for dysphagia treatment in tracheotomized stroke patients: a randomized controlled trial. Intensive Care Med. 2015 Sep;41(9):1629-37. doi: 10.1007/s00134-015-3897-8. Epub 2015 Jun 13. PMID 26077087